CLINICAL TRIAL: NCT04727268
Title: Genotype-phenotype Correlation in Junctional Epidermolysis Bullosa
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: Dystrophic Epidermolysis Bullosa Research Association (DEBRA) (Unknown); University of Birmingham (Other)
Responsible Party: Principal Investigator, Dr David Wen, Dermatology Fellow, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK7326
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Junctional Epidermolysis Bullosa; Laryngo Onycho Cutaneous Syndrome
Keywords: Open access database; Junctional Epidermolysis Bullosa; Genotype phenotype correlation
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional; Laryngo onycho cutaneous syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Retrospective data regarding genetic information will be collected from participants' medical records.
  Deep phenotyping of participants will also be completed.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No interventions present in this study.

SUMMARY:
This study will collect genetic and clinical information of junctional epidermolysis bullosa (JEB) patients. Computer analysis will be performed on genetic mutations found in these patients and this will be correlated with their clinical characteristics.

DETAILED DESCRIPTION:
Junctional epidermolysis bullosa (JEB) is a rare genetic skin disease where genetic defects in skin proteins result in extensive blistering in response to mild mechanical stress. Patients are often affected at birth or from early childhood, and suffer from varying degrees of severity depending on the specific mutations that they have and the proteins that are affected. This ranges from severe widespread blistering and death within the first few years of life, to minimal localised blistering and survival to adulthood. Diagnosis is confirmed by genetic testing, and this is often used to predict the likely clinical course. However, it is not always straightforward to make accurate predictions from genetic information, as our understanding of these proteins and mutations at the molecular level is currently incomplete.

The main aim of this project is to systematically collect genetic and clinical data of junctional epidermolysis bullosa (JEB) patients and to explore whether there are any relationships between participants' genetic defects and the severity of disease. This will help in establishing links between genetic defects and clinical characteristics, which is essential for accurate prognostication, genetic counselling and prenatal diagnosis.

This study will also aim to develop pipelines for analysis of how mutations may affect corresponding protein structure and function using computer prediction tools. This will improve our understanding of how these proteins function, and could partly explain the variation in disease severity of patients with this condition. It could also lead to identification of important regions of the protein, which could be investigated further in subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

Adults and children with a diagnosis of JEB or LOC syndrome, which has been confirmed with genetic testing. A mutation is present in one of the following genes: LAMA3, LAMB3, LAMC2 or COL17A1.

Current JEB patients, or JEB patients within the last 5 years who have used the EB service at Solihull hospital or Birmingham Women's and Children's Hospital. This includes patients who are living and also those who passed away in the last 5 years (eg from severe JEB).

Exclusion Criteria:

Adult patients who are unable to give informed consent. Child patients who do not assent and/ or have no one appropriate who can consent on their behalf.

Persons who might not adequately understand verbal explanations or written information given in English.

Ages: 0 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with JEB, confirmed through genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Genotype and phenotype data collection | 6 months
  The primary objective is to systematically collect genetic and clinical data of junctional epidermolysis bullosa (JEB) patients and to explore whether there are any relationships between participants' genetic defects and the severity of disease.

SECONDARY OUTCOMES:
Bioinformatic analysis | 10 months
  Development of a pipeline for bioinformatic analysis of variants

CONTACTS AND LOCATIONS:
Locations (1):
- Solihull Hospital, Solihull, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once data collection and analysis has been completed, anonymised data regarding genotype and phenotype will be presented at scientific meetings and publised in journals and / or postgraduates theses.

REFERENCES:
- [Background] Has C, Bauer JW, Bodemer C, Bolling MC, Bruckner-Tuderman L, Diem A, Fine JD, Heagerty A, Hovnanian A, Marinkovich MP, Martinez AE, McGrath JA, Moss C, Murrell DF, Palisson F, Schwieger-Briel A, Sprecher E, Tamai K, Uitto J, Woodley DT, Zambruno G, Mellerio JE. Consensus reclassification of inherited epidermolysis bullosa and other disorders with skin fragility. Br J Dermatol. 2020 Oct;183(4):614-627. doi: 10.1111/bjd.18921. Epub 2020 Mar 11. PMID 32017015
- [Background] Bardhan A, Bruckner-Tuderman L, Chapple ILC, Fine JD, Harper N, Has C, Magin TM, Marinkovich MP, Marshall JF, McGrath JA, Mellerio JE, Polson R, Heagerty AH. Epidermolysis bullosa. Nat Rev Dis Primers. 2020 Sep 24;6(1):78. doi: 10.1038/s41572-020-0210-0. PMID 32973163